CLINICAL TRIAL: NCT03437226
Title: Repetitive Levosimendan Infusion for Patients With Advanced Chronic Heart Failure
Acronym: LeoDOR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Gerhard Pölzl (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor-Investigator, Dr. Gerhard Pölzl, Univ. Prof. Dr. med., Medical University Innsbruck
Organization: Medical University Innsbruck (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LeoDOR2017
Record Dates: First submitted 2017-10-09; First posted 2018-02-19 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure
Keywords: Heart Failure, Levosimendan
MeSH Terms: conditions — Heart Failure | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levosimendan Arm (Experimental): Patients receive 6 or 24 hours infusion depending on the site. Levosimendan 2.5 MG/M 6h infusion group: 0,2 μg/kg/min 7 times (day 0, 14, 28, 42, 56, 70, 84) Levosimendan 24h infusion group: 0,1 μg/kg/min 5 times (day 0, 21,42,63,84) Levosimendan
  Interventions: Drug: Levosimendan 2.5 MG/ML
- Placebo Arm (Placebo Comparator): Patients receive 6 or 24 hours infusion depending on the site. 6h infusion group: 0,2 μg/kg/min 7 times (day 0, 14, 28, 42, 56, 70, 84) Placebo 24h infusion group: 0,1 μg/kg/min 5 times (day 0, 21,42,63,84) Placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Levosimendan 2.5 MG/ML — Levosimendan Arm: 1 x 5 ml (1 vial) of levosimendan infusion concentrate is added to one 250 ml infusion bag of 5% glucose or 0.9% NaCl in diabetic patients.
  Other Names: Simdax, Orion Pharma, Espoo, Finland
  Arms: Levosimendan Arm
Drug: Placebos — Placebo Arm: 1 x 5 ml (1 vial) of placebo levosimendan infusion concentrate is added to one 250 ml infusion bag of 5% glucose or 0.9% NaCl in diabetic patients.
  Other Names: Placebo Levosimendan infusion concentrate
  Arms: Placebo Arm

SUMMARY:
Repetitive levosimendan infusions for patients with advanced chronic heart failure (LeoDOR) A randomised, double-blind, placebo-controlled multicentre study with parallel group design.

Mortality and rehospitalisation rates are high in the vulnerable phase following heart failure hospitalisation. Previous studies suggest that these events can be reduced by repeat infusions of levosimendan in patients with advanced heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Written, signed and dated informed consent.
2. Male and female patients over 18 years of age.
3. Women of childbearing potential must have a monthly negative pregnancy test and must refrain from breastfeeding. Women who are postmenopausal (1 year since last menstrual cycle), surgically sterilised or who have undergone a hysterectomy are considered not to be of childbearing potential.
4. CHF diagnosed at least 6 months before screening and treated with individually optimised long-term oral treatment for the last month, unless not tolerated (e.g., ACE-inhibitor or AT II blocker, beta-blocker, mineralocorticoid receptor antagonist, angiotensin II receptor blocker neprilysin inhibitor [ARNI] and with devices [e.g., CRT/ICD], as needed).
5. Left ventricular ejection fraction less than or equal to 30% as assessed by echocardiography, radionuclide ventriculography or contrast angiography within the index hospitalisation.
6. Currently hospitalised for decompensated HF requiring i.v. diuretics, or i.v. vasodilators, or i.v. inotropic therapy, or their combination.
7. Previous hospitalisation or visit to outpatient clinic requiring i.v. diuretics, i.v. vasodilators, or i.v. inotropic therapy, or their combination for acute decompensated HF within 12 months before the current hospitalisation.
8. NT-proBNP level after recompensation of more or equal 2500 ng/L (BNP more or equal 900 ng/L) and/or NYHA class III or IV at study entry

Exclusion Criteria:

1. Severe obstruction of ventricular outflow tracts such as haemodynamically significant uncorrected primary valve disease or hypertrophic cardiomyopathy or impaired ventricular filling such as restrictive cardiomyopathy.
2. Predominantly right heart failure a/o severe tricuspid regurgitation
3. Cardiac surgery or coronary angioplasty within 30 days before study drug initiation.
4. Acute coronary syndrome within 30 days before study drug initiation.
5. Patients who are scheduled for cardiac surgery or angioplasty in the next 3 months
6. History of torsades de pointes
7. Stroke or transient ischaemic attack (TIA) within 3 months before study drug initiation
8. Systolic blood pressure less than 90 mmHg at baseline
9. Heart rate 120 bpm or greater at baseline
10. Serum potassium less than 3.5 mmol/l before study drug initiation.
11. Severe renal insufficiency (estimated glomerular filtration rate (eGFR) <30 ml/min/1.73m2)
12. Anaemia (haemoglobin < 10 g/dl)
13. Significant hepatic impairment at the discretion of the investigator.
14. Hypersensitivity to levosimendan
15. Other serious diseases limiting life expectancy considerably (e.g. end-stage cancer, end-stage lung disease)
16. Participation in a clinical trial with any experimental treatment within 30 days prior to screening or previous participation in the present study
17. Administration of levosimendan within 14 days prior the study drug initiation, the first study drug application has to be postponed for at least 14 days after the end of this premedication
18. Suspected non-compliance
19. Pregnant woman and nursing mother
20. Failure to use highly-effective (Pearl Index lower than 1%) contraceptive methods.
21. Person with any kind of dependency on the investigator
22. Person held in an institution by legal or official order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2018-03-08 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to death, high-urgent heart transplantation or ventricular assist device (VAD), time to non-fatal HF event | From baseline (day 1) up to Follow-up 2 (day 180)
  Time to event in days, from baseline visit (day 1) up to Follow-up 2 (day 180)
Change in NT-proBNP | Change from Baseline NT-proBNP (day 1) to Follow-up 1 (day 90)
  pg/ml

SECONDARY OUTCOMES:
Change in functional status and symptoms via KCCQ (Combined Outcome measurement) | From baseline (day 1) up to day 98 (FUP 1)
  KCCQ (Kansas City Cardiomyopathy Questionnaire) The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life.
Change in functional status and symptoms via PGA (Combined Outcome measurement) | From baseline (day 1) up to day 98 (FUP 1)
  PGA (Patient's global assessment)
Change in functional status and symptoms via EQ-5D-5L (Combined Outcome measurement) | From baseline (day 1) up to day 98 (FUP 1)
  EQ-5D-5L VAS is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal visual analogue scale
cumulative number of: days alive out of hospital (Combined Outcome measurement) | From baseline (day 1) up to day 180 (FUP 2)
  Counted in days
cumulative number of: non-fatal HF events (Combined Outcome measurement) | From baseline (day 1) up to day 180 (FUP 2)
  Counted in events
cumulative number of: hospital admissions (Combined Outcome measurement) | From baseline (day 1) up to day 180 (FUP 2)
  counted in numbers
death | From baseline (day 1) to day 180 (FUP 2)
  Number of participants died within the defined time points
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | From baseline (day 1) to day 180 (FUP 2)
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 counted in numbers

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No